CLINICAL TRIAL: NCT05755854
Title: Allogeneic γ9δ2 T Cells for the Treatment of Recurrent Hematologic Tumors After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Allogeneic γ9δ2 T Cells Treatment of Recurrent Hematologic Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Xiaoyu Zhu, Director of Hematology Department, Anhui Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QH10103-M-01（0）
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Hematologic Diseases
Keywords: Recurrent hematologic tumors; Allogenic γδT Cell
MeSH Terms: conditions — Hematologic Diseases | interventions — fludarabine; fludarabine phosphate; Injections; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with recurrent hematologic tumors after allogeneic hematopoietic stem cell transplantation (Experimental): A conditional chemotherapy regimen of fludarabine and cyclophosphamide will be administered, zoredronic acid depending on the patient's status, followed by investigational therapy, allogeneic γ9δ2 T Cells
  Interventions: Biological: allogeneic γ9δ2 T Cells; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Zoredronic acid

INTERVENTIONS:
Biological: allogeneic γ9δ2 T Cells — dose escalation (3+3) : dose 1 (5 × 10^7cells/kg) ,dose 2 (1 × 10^8 cells/kg) ,dose 3 (2 × 10^8cells/kg)
Drug: Fludarabine — Intravenous fludarabine on days-5 and -4,the infusion dose is adjusted according to the subject's condition
  Other Names: Fludarabine Phosphate for Injection
Drug: Cyclophosphamide — Intravenous cyclophosphamide on days -5、-4、and -3, the infusion dose is adjusted according to the subject's condition
  Other Names: Cyclophosphamide for Injection
Drug: Zoredronic acid — Intravenous zoredronic acid 50ug/kg 24 hours before cell infusion（or according to the dosage of the instruction）（If applicable）

SUMMARY:
This is an open single-arm clinical study aimed at evaluating the safety and tolerance of allogeneic γ9δ2 T cell injection in the treatment of patients with recurrent hematologic tumors after allogeneic hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
To evaluate the safety and in vivo dynamics of allogeneic γ9δ2 T cell in the treatment of recurrent hematologic tumors after allogeneic hematopoietic stem cell transplantation patients, and to explore the appropriate therapeutic dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12-65 (inclusive)；
2. Patients with recurrent hematologic tumors after allogeneic hematopoietic stem cell transplantation；
3. Basically normal liver and kidney function (as demonstrated by the following laboratory tests prior to initial γ9δ2 T cell therapy)

   * Alanine transaminase/aspartate transaminase < 2.5×ULN；
   * serum creatinine < 1.5×ULN；
   * total bilirubin level < 1.5×ULN；
4. No obvious hereditary disease;
5. Normal cardiac function, cardiac ejection index above 55%;
6. Women of reproductive age (15 to 49 years) must undergo a pregnancy test within 7 days before starting treatment and the result is negative, and use contraception during the clinical trial period and within 3 months after the last cell transfusion;
7. Sign informed consent.

Exclusion Criteria:

1. Patients with simple extramedullary recurrence;
2. Pregnant and lactating women;
3. Organ failure;

   * Heart: Ⅲ level and Ⅳ level;
   * Liver: reach the grade C Child - Turcotte liver function;
   * Kidney, renal failure and uremia period;
   * Lung: symptoms of severe respiratory failure;
   * Brain: consciousness disorder.
4. Patients with a history of solid organ transplantation;
5. Uncontrollable infectious diseases or other serious diseases, including but not limited to infections (such as HIV positive), congestive heart failure, unstable angina, arrhythmia, psychosis, or restricted social circumstances or those that the attending physician considers to pose unpredictable risks;
6. Patients with systemic autoimmune diseases or primary immunodeficiency;
7. Patients with allergic constitution;
8. Use of systemic steroid drugs;
9. Chronic diseases requiring the use of immunological agents or hormone herapy;
10. Prior treatment with any other immune cells;
11. Participated in similar clinical trials within 30 days;
12. Received radiation therapy within 4 weeks from the time of enrollment;
13. Researchers don't think clinical trials are appropriate for other reasons.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | 12 months
  AE is defined as any adverse medical event from the date of leukapheresis to 12 months after allogeneic γ9δ2 T cells infusion. Among them, cytokine release syndrome (CRS) and immune cell-associated neurotoxicity syndrome (ICANS) were graded according to American Society for Transplantation and Cellular Therapy (ASTCT) criteria, graft-versushost disease (GVHD) according to criteria defined by the Mount Sinai Acute GVHD International Consortium. Other AEs were graded according to common terminology criteria for adverse events (CTCAE) v5.0
Incidence of Dose-Limiting Toxicities (DLTs) | First infusion date of allogeneic γ9δ2 T cells to 14 days end cell infusion
  DLT was defined as allogeneic γ9δ2 T Cells-related events with onset within first 14 days following infusion:
  The development of Grade (G) III-IV acute GVHD according to the Mount Sinai Acute GVHD International Consortium criteria; The development of G3 or higher grade CRS lasting > 2 weeks; Any allogeneic γ9δ2 T cells-related AE requiring intubation; All G4 non-hematologic toxicities. Symptoms of GVHD include but are not limited to skin rash, enterocolitis with diarrhea, liver dysfunction with jaundice, fever, weight loss, etc.
Maximum tolerated dose (MTD) | 14 days
  MTD is defined as the highest dose level of less than or equal to 2 DLT among the 6 subjects finally determined.
Recommended phase 2 dose (RP2D) | 14 days
  The recommended dose for phase 2 was determined through phase 1 study

SECONDARY OUTCOMES:
Overall Survival (OS) | 12 months
  OS is defined as the time from allogeneic γ9δ2 T cells infusion to the date of death. Subjects who have not died by the analysis data cutoff date will be censored at their last contact date.
Progression Free Survival (PFS) | 12 months
  PFS is defined as the time from the allogeneic γ9δ2 T cells infusion date to the date of disease progression assessed by investigators assessment, or death any cause. Participants not meeting the criteria for progression by the analysis data cutoff date were censored at their last evaluable disease assessment date.
Pharmacokinetics: Persistence of the allogeneic γ9δ2 T cells | 14 days
  Persistence of the allogeneic γ9δ2 T cells assessed by number in peripheral blood.
Pharmacodynamics: Peak level of cytokines in serum | 14 days
  The cytokines mainly include interleukin-2 (IL-2 ), IL-6, IL-8, IL-10, tumor necrosis factor-α (TNF-α) etc. Peak was defined as the maximum post-baseline level of the cytokine.

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Xiaoyu, Ph.D, Principal Investigator — Director of Hematology Department, Anhui Provincial Hospital
Locations (1):
- Anhui Provincial Hospital, Hefei, Anhui, China